CLINICAL TRIAL: NCT06476327
Title: The Effects of Robot-Assisted Gait Training Concurrent With Self-Observation Training on Balance, Gait, Cognitive Function in Stroke
Brief Title: Robot-Assisted Gait Training With Self-Observation in Stroke Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYU 2024-05-017
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: stroke; gait; cognitive function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental 1 group (Active Comparator): Robot-Assisted Gait with Self-Observation
  Interventions: Behavioral: experimental 1 group
- experimental 2 group (Active Comparator): Robot-Assisted Gait
  Interventions: Behavioral: experimental 2 group

INTERVENTIONS:
Behavioral: experimental 1 group — A camera is installed on the walker used in the training, and the recorded video is mirrored in real-time to a tablet computer. Participants can view this video through smart glasses connected to the tablet computer. A glasses strap will be used to secure the glasses, ensuring there is no interference with walking.
  Participants will undergo a total of 20 training sessions, five times a week for four weeks, with each session lasting 30 minutes. Participants will have a 4-minute break during the 30-minute gait training session.
  Participants will be given a period to adapt to wearing the robot, and after that, the intervention will be conducted based on each participant's individual abilities and adaptation.
  Arms: experimental 1 group
Behavioral: experimental 2 group — Participants will undergo a total of 20 training sessions, five times a week for four weeks, with each session lasting 30 minutes. Participants will have a 4-minute break during the 30-minute gait training session.
  Participants will be given a period to adapt to wearing the robot, and after that, the intervention will be conducted based on each participant's individual abilities and adaptation.
  Arms: experimental 2 group

SUMMARY:
The aim of this study is to investigate the effects of robot-assisted gait training Concurrent with self-observation training on balance, gait, and cognitive function in stroke participants. The main question it aims to answer is:

Does robot-assisted gait training combined with self-observation improve balance abilities in stroke participants?

Participants will be

Group 1 Perform robot-assisted gait training combined with self-observation five times a week for four weeks.

Group 2 Perform robot-assisted gait training five times a week for four weeks.

All groups perform for 30 minutes per session.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have had a stroke for more than 6 months but less than 1 year
* Functional Ambulation Category (FAC) ≥ 2
* Able to walk 10 meters independently with or without an assistive device
* Participants eligible for application of the robot (ANGEL LEGS M20, Anger Robotics)

Exclusion Criteria:

* Inability to wear the robot due to open wounds or skin conditions
* Severe cognitive impairment (MMSE-K < 10) or significant difficulty in communication due to language disorders
* Spasticity of the paralyzed limb with a Modified Ashworth Scale (MAS) ≥ 2
* High risk of fractures, such as osteoporosis
* Severe cardiovascular or pulmonary diseases
* Neurological disorders affecting gait function, such as Parkinson's disease or multiple sclerosis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Balance ability | from enrollment to the end of treatment at 4 weeks
  - Timed up and go test (TUG)
  Participants sit on a chair with armrests, rise upon hearing a starting signal, walk 3 meters, return, and sit back down. The speed of this task is measured. Participants may use usual walking aids (cane or walker) but should not receive physical assistance.
  - Functional Reach Test (FRT)
  Participants stand against a wall with feet fixed vertically, arms raised to 90 degrees, reaching forward as far as possible while measuring the distance (in cm) from the tip of the third metacarpal bone.
Gait ability | from enrollment to the end of treatment at 4 weeks
  -10 meter walking test (10MWT)
  The walking speed is calculated by measuring the time (in seconds) takes for the subject to walk 10 meters. Instructed to walk a total of 14 meters at maximum speed, excluding the first 2 meters and the last 2 meters to account for acceleration and deceleration phases. Participants may use personal walking aids (cane, walker, etc.).
  -GAITRite system (CIR Systems Inc., Franklin, New Jersey, USA)
  Participants pass over an electronic gait mat to computationally measure temporal and spatial walking variables.

SECONDARY OUTCOMES:
Cognitive ability | from enrollment to the end of treatment at 4 weeks
  - Mini-Mental Status Examination-Korea, (MMSE-K)
  Consists of memory, recall ability, attention, language skills, numerical ability, and constructional ability.
  Memory has 10 points, registration has 3 points, attention and calculation have 5 points, recall has 3 points, language function has 7 points, and comprehension and judgment have 2 points, totaling six areas and twelve items

CONTACTS AND LOCATIONS:
Locations (1):
- Chungdam hospital, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No